CLINICAL TRIAL: NCT05891938
Title: Effects of Hydrogen Gas Inhalation on Community-Dwelling Adults of Various Ages: A Single-Arm, Open-Label, Prospective Clinical Trial
Brief Title: Effects of Hydrogen Gas Inhalation on Adults of Various Ages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Kyu Jae Lee, Professor, Wonju Severance Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EMB-2023-01
Record Dates: First submitted 2023-05-01; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: Before and after of treatment in single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single group treatment
  Interventions: Other: H2 gas inhalation

INTERVENTIONS:
Other: H2 gas inhalation — H2 gas inhalation treatment for 4 weeks in on community dwelling adults of various ages

SUMMARY:
Herein, investigated the effects of 4 weeks of H2 gas inhalation on community-dwelling adults of various ages.

DETAILED DESCRIPTION:
Molecular hydrogen (H2) is a versatile therapeutic agent. H2 gas inhalation is reportedly safe and has a positive impact on a range of illnesses, including Alzheimer's disease (AD). Herein, investigated the effects of 4 weeks of H2 gas inhalation on community-dwelling adults of various ages. Fifty-four participants including those dropped out (5%) were screened and enrolled. The selected participants were treated as a single group without randomization. Evaluated the association between total and differential white blood cell (WBC) counts and AD risk at individual levels after 4 weeks of H2 gas inhalation treatment. Furthermore, evaluation of dementia-related biomarkers such as beta-site APP cleaving enzyme 1 (BACE-1), amyloid beta (Aβ), brain-derived neurotrophic factor (BDNF), vascular endothelial growth factor A (VEGF-A), T-tau, monocyte chemotactic protein-1 (MCP-1), and inflammatory cytokines (interleukin-6).

ELIGIBILITY:
Inclusion

* Age ranges 40-70 years
* Healthy participants
* Patients who are willing or able to follow the doctor's instructions
* Fully understand the purpose and procedure of this clinical trial

Exclusion Criteria

* Participants excluded those who have any disease
* Pregnant and lactating women

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Measurement of white blood cell and its differential counts such as neutrophils (%), basophils (%) | 4 weeks
  4 weeks treatment of H2 gas inhalation in community dwelling adults of various ages
Measurement of oxidative stress markers such as reactive oxygen species (µM), and nitric oxide (µM) | 4 weeks
  4 weeks treatment of H2 gas inhalation in community dwelling adults of various ages

SECONDARY OUTCOMES:
Measurement of dementia biomarkers such as brain-derived neurotrophic factor (BDNF ng/mL) | 4 weeks
  4 weeks treatment of H2 gas treatment
Measurement of dementia biomarkers such as brain-derived neurotrophic factor amyloid beta (Aβ (pg/mL)) | 4 weeks
  4 weeks treatment of H2 gas treatment
Measurement of inflammatory markers such as interleukin 6 (pg/mL) | 4 weeks
  4 weeks treatment of H2 gas treatment

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Kyu Jae Lee, Ph.D., Study Chair — Wonju College of Medicine
Locations (2):
- South Korea (2):
  - Wonju College of Medicine, Wŏnju, Ganwon-do
  - Wonju Severance Christian Hospital, Wŏnju, Gwando

IPD SHARING:
Plan to Share IPD: No